CLINICAL TRIAL: NCT05287750
Title: Brain Diseases on 7.0T Magnetic Resonance Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Director and Clinical Professor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Brain Diseases-ChinaPLAGH
Record Dates: First submitted 2022-01-07; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Brain Tumor; MRI; Cerebrovascular Disease
Keywords: Brain tumor; Cerebrovascular disease; MRI; Ultra high field
MeSH Terms: conditions — Brain Neoplasms; Cerebrovascular Disorders | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — Patients recruited will receive Magnetic resonance imaging.

SUMMARY:
This clinical trial studies the use of 7-Tesla (7T)and 3T magnetic resonance imaging (MRI) in detecting brain diseases. 7T MRI has increased detection sensitivity, including more accurate lesion delineation, higher inter-rater agreement. Diagnostic procedures such as 7T MRI may help ultimately improved diagnostic and therapies confidence to inform decision making than standard 3T MRI.

DETAILED DESCRIPTION:
7T MRI increased detection sensitivity, attain superior anatomic resolution, higher spatial and spectral specificity of advanced quantitative techniques, and shorter scan times than 3T MRI. When applied clinically, these benefits translate to increased detection sensitivity, and ultimately improved diagnostic and therapies confidence to inform decision making. This study aim to detect the image characteristics and diagnostic accuracy of brain diseases on 7T MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 and ≤80
* Having brain diseases (eg: brain tumor, cerebrovascular diseases)
* Having no contraindications against MRI or intravenous contrast agent administration
* Clinically stable

Exclusion Criteria:

* Age<18 or >80
* Pregnancy and other contraindication to MRI scan
* Informed consent not obtained

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
the correspondence between brain tumor cells found in the biopsies and region of interest(ROI) signal intension on the 7T MRI scan and 3T MRI scan | within a month after biopsy
  Pathological assessment of biopsy material compared with the lesion's contrast-enhancement signal intension to normal brain white mater on 7T MRI and 3T MRI
The visibility of white matter tracts on 7T MRI | within a month after biopsy
  Visualization of white matter tracts will be done with the use of diffusion tensor imaging (DTI) on 7T MRI and measuring the mean diffusivity (MD) value on Post-processing workstation ,and analysis the correlation between these values and pathological.

SECONDARY OUTCOMES:
The correlation between the ROI's signal intension on 7T MRI scan and the KPS in 1 month after operation | within a month after biopsy
  The correlation analysis between the T1 contrast-enchanced signal intension, Regional cerebral blood flow on 7T MRI (clinical sequence and perfusion) scan and the KPS in 1 month after operation
The visibility of white matter tracts on 7T MRI and 3T MRI | Six months after the biopsy
  Visualization of white matter tracts will be done with the use of diffusion tensor imaging (DTI) on 7T MRI and 3T MRI. and analysis the difference of the mean diffusivity (MD) value between 7.0T MRI and 3.0T MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

REFERENCES:
- [Derived] Duan Q, Lyu J, Liu Z, Hao F, Li R, Liu S, Hao X, Li J, Bian X, Duan C, Wang S, Wang W, Wang R, Duan L, Lou X. Noninvasive Assessment of the Risk Features of Hemorrhage in Moyamoya Disease Using 7T MRI. Neurology. 2025 Jun 10;104(11):e213617. doi: 10.1212/WNL.0000000000213617. Epub 2025 May 21. PMID 40397837
- [Derived] Duan C, Bian X, Cheng K, Lyu J, Xiong Y, Xiao S, Wang X, Duan Q, Li C, Huang J, Hu J, Wang ZJ, Zhou X, Lou X. Synthesized 7T MPRAGE From 3T MPRAGE Using Generative Adversarial Network and Validation in Clinical Brain Imaging: A Feasibility Study. J Magn Reson Imaging. 2024 May;59(5):1620-1629. doi: 10.1002/jmri.28944. Epub 2023 Aug 9. PMID 37559435